CLINICAL TRIAL: NCT04302805
Title: rATG Versus rATG Combined With IVIG Induction Immunosuppression in HLA Incompatible Transplantation
Brief Title: rATG Versus rATG Combined With Intravenous Immunoglobulin (IVIG) Induction Immunosuppression in HLA Incompatible Transplantation (INHIBIT)
Acronym: INHIBIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Ondřej Viklický, M.D., Ph.D., Head of Department of Nephrology and Transplant Center, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Eudra CT: 2019-003723-37
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplantation
Keywords: Antibody-mediated rejection; Intravenous immunoglobulin; Rabbit Anti-thymocyte Globulin; Donor specific antibodies
MeSH Terms: interventions — Immunoglobulins, Intravenous; thymoglobulin; Plasma Exchange

STUDY DESIGN:
Intervention Model Description: The present study is a prospective randomized single-centre open-label two-arm Phase III.b non-inferiority clinical trial. This trial aims to prove similar efficacy of PE/rATG and PE/rATG/IVIG (centre standard of care) induction regimens to prevent biopsy proven antibody-mediated changes and TCMR as composite endpoint within 12 months after HLA incompatible kidney transplantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PE/rATG (Placebo Comparator): Study participants will undergo therapeutic plasma exchange (PE, 1 plasma volume) before the transplant surgery and receive rATG (Thymoglobuline®) induction (1.5 mg/kg intraoperatively and 1 mg/kg when possible daily within first week up to cumulative dose 5-7 mg/kg).
  Interventions: Drug: Thymoglobulin; Other: Plasma Exchange
- PE/rATG/IVIG (Active Comparator): Study participants will undergo therapeutic plasma exchange (PE, 1 plasma volume) before the transplant surgery and receive rATG (Thymoglobuline®) induction (1.5 mg/kg intraoperatively and 1 mg/kg when possible daily within first week up to cumulative dose 5-7 mg/kg) and IVIG 0.5g/kg intravenous infusions, on 1st, 3rd and 5th postoperative day. This is a center standard of care regimen.
  Interventions: Drug: Privigen; Drug: Thymoglobulin; Other: Plasma Exchange

INTERVENTIONS:
Drug: Privigen — Patients randomized to PE/rATG/IVIG group will receive IVIG 0.5g/kg infusions, on 1st, 3rd and 5th postoperative day.
  Other Names: IVIG; Kiovig
  Arms: PE/rATG/IVIG
Drug: Thymoglobulin — All patients will receive 1.5 mg/kg intraoperatively and 1 mg/kg when possible daily within first week up to cumulative dose 5-7 mg/kg.
  Other Names: rATG
Other: Plasma Exchange — All patient will undergo Plasma Exchange before transplantation.
  Other Names: PE

SUMMARY:
This study aims to prove similar efficacy of PE/rATG (intervention) and PE/rATG/IVIG (centre standard of care) induction regimens to prevent biopsy proven antibody-mediated changes and TCMR as composite endpoint within 12 months after HLA incompatible kidney transplantation.

DETAILED DESCRIPTION:
There have been no published clinical studies evaluating rATG/IVIG induction protocol in comparison with rATG alone in defined cohort of HLA incompatible kidney transplant recipients. Prescribing IVIG in management of prevention of transplant rejection is considered off-label use, however IVIG remains part of induction protocols in many transplant centres. IVIG therapy is demanding due to high cost and limited resources of these human origin products. Trial participants will be end-stage renal disease (ESRD) patients listed for deceased donor / living donor kidney transplantation with anti HLA antibody screening performed within 12 months before transplantation and with last DSA 1 000 - 5 000 Mean Fluorescence Intensity (MFI) and negative CDC (Complement-dependent cytotoxicity crossmatch test) prior to transplantation. Participants will be randomized into one of the treatment groups (PE/PP(Plasmapheresis) + rATG + IVIG, PE/PP + rATG) and as a primary outcome a composite endpoint defined as occurrence of antibody- or T-cell mediated rejection within 12 months after transplantation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Primary deceased donor or living donor kidney transplantation (first transplantation or re-transplantation)
* Recipient age ≥ 18 years and < 70 years
* Donor age < 70 years
* Written Informed Consent and Consent for Processing Personal Data
* Last anti-HLA screening no longer than 12 months with positive results
* MFI DSA 1 000 - 5 000 (anti-HLA A, B, DR), MFI DSA 1000-15000 for anti DQ when available at randomization)

Exclusion Criteria:

* Combined kidney transplantation with another organ
* Immunosuppressive therapy up to 6 months before transplantation
* AB0i (AB0 incompatible) transplantation
* Women in childbearing potential without adequate contraception
* HIV positivity
* Leukopenia < 3 000, thrombocytopenia < 75 000
* Tuberculosis history
* Anti-HCV (Hepatitis C Virus) positivity, HBsAg (Hepatitis B Surface Antigen) positivity or HBV (Hepatitis B Virus) DNA positivity
* DSA (anti A, B, DR) measured by Luminex with MFI > 5 000 known at screening prior to transplant, anti DQ > 15000 if known
* FACS (flow-cytometry) T and B crossmatch positivity known at screening prior to transplant
* Positive CDC prior to transplantation
* Planned PP/PE and RTX (Rituximab) treatment post-transplant
* Advanced liver disease (Child-Pugh C or laboratory values of ALT or AST more than 3 times upper limit of normal range)
* Pregnancy, breastfeeding
* Study medication is contraindicated according to the SmPC
* Patient is enrolled in other clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Combined endpoint defined as biopsy proven antibody mediated changes (Banff 2017, Category 2) and/or TCMR (Banff 2017, Category 4) regardless the biopsy indication (for cause or protocol biopsy) in HLAi (HLA incompatible)kidney transplantation | 12 months
  Number of biopsy-confirmed rejections

SECONDARY OUTCOMES:
Incidence of active antibody-mediated rejection (ABMR) lesions within 12 months post-transplantation | 12 months
  Number of active active antibody-mediated rejection (ABMR) lesions within 12 months post-transplantation
Time to active antibody-mediated rejection (ABMR) within 12 months post-transplantation | 12 months
  Time to active antibody-mediated rejection (ABMR) occurrence in months
Incidence of chronic active antibody-mediated rejection (ABMR) and C4d staining without evidence of rejection in protocol biopsies at Month 3 and Month 12 | 3 and 12 months
  Number of chronic active antibody-mediated rejection (ABMR) and C4d staining without evidence of rejection in protocol biopsies at Month 3 and Month 12
Incidence of transplant glomerulopathy (TG) in protocol biopsies at Month 3 and Month 12 | 3 and 12 months
  Number of biopsies with transplant glomerulopathy
Incidence of acute T-cell mediated rejection (TCMR) and chronic active TCMR in protocol biopsies at Month 3 and Month 12 post-transplantation | 3 and 12 months
  Number of acute T-cell mediated rejection (TCMR) and chronic active TCMR in protocol biopsies at Month 3 and Month 12
Estimated glomerular filtration rate (eGFR) at Month 3, Month 6 and Month 12 | 3, 6 and 12 months
  Estimated glomerular filtration rate (eGFR) will be assessed at all study visits by CKD-EPI formula.
Measured proteinuria and albuminuria at Month 3, Month 6 and Month 12 | 3, 6 and 12 months
  Proteinuria is defined as ≥ 1 g/l and albuminuria as albumin/creatinine ratio > 3 mg/mmol.
Donor specific antibodies (DSA) at Month 3, Month 6 and Month12 | 3, 6 and 12 months
  Specification of antibodies directed at HLA class I and class II will be performed by LUMINEX method (solid phase assay).
De novo donor specific antibodies (DSA) at Month 3, Month 6 and Month 12 | 3, 6 and 12 months
  Specification of antibodies directed at HLA class I and class II will be performed by LUMINEX method (solid phase assay).
Mortality rate within 12 months post-transplantation | 12 months
  Number of deaths by any cause anytime during the trial.
Graft survival (rate of graft loss) within 12 months post transplantation | 12 months
  Number graft of graft failures within 12 months
Incidence of metabolic, malignant and cardiovascular co-morbidities | 12 months
  Number of metabolic, malignant and cardiovascular co-morbidities
Incidence of viral and bacterial complications | 12 months
  Number of viral and bacterial complications
Incidence of BK Virus (BKV), Cytomegalovirus (CMV) and Epstein-Barr Virus (EBV) replications detected by PCR (polymerase chain reaction) at Month 3, Month 6 and Month 12 | 3, 6 and 12 months
  Number of patients with PCR (polymerase chain reaction) positive BK Virus (BKV), Cytomegalovirus (CMV) and Epstein-Barr Virus (EBV) replications
Incidence of study treatment discontinuation | 12 months
  Cessation of trial medication treatment either by the clinician or by the participant himself/herself.
Incidence of molecular rejection in the 12-month protocol biopsies | 12 months
  Number of molecular rejection cases evaluated by the Molecular Microscope Diagnostic System (MMDx) in the 12-month protocol biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Viklicky, Prof., Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viklicky O, Zahradka I, Mares J, Slatinska J, Parikova A, Petr V, Roder M, Jaklova K, Osickova K, Janousek L, Hruba P. 12-Month Outcomes of a Prospective Randomized Trial Investigating Effects of IVIG on Top of rATG Versus rATG Alone in Pre-Sensitized Kidney Transplant Recipients: The INHIBIT Study. Transpl Int. 2025 May 19;38:14312. doi: 10.3389/ti.2025.14312. eCollection 2025. PMID 40458542